CLINICAL TRIAL: NCT00626730
Title: Adjuvant Postoperative High-Dose Radiotherapy for Atypical and Malignant Meningioma: a Phase-II and Observation Study
Brief Title: Radiation Therapy in Treating Patients Who Have Undergone Surgery for Newly Diagnosed Grade II or Grade III Meningioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: EORTC-22042-26042; EORTC-22042; EORTC-26042; 2005-005551-18 (EudraCT Number)
Record Dates: First submitted 2008-02-28; First posted 2008-02-29 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult grade II meningioma; adult grade III meningioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Meningioma | interventions — Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving high-dose radiation therapy after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying radiation therapy to see how well it works in treating patients who have undergone surgery for newly diagnosed grade II or grade III meningioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the impact of high-dose radiotherapy (RT) on progression-free survival (PFS), treatment tolerance, and post-treatment global cognitive functioning in patients with atypical (WHO grade II) or malignant ( WHO grade III) meningioma.

OUTLINE: Patients with grade II disease are stratified according to resection status (complete excision [Simpson's stages 1-3] vs incomplete excision [Simpson's stages 4-5]) and participate in a phase II study. These patients are assigned to 1 of 2 treatment groups according to Simpson staging. Only data from these patients is analyzed with respect to the progression-free survival endpoint. Patients with grade III disease are treated in group 1 or 2 according to Simpson staging (as patients with grade II disease). After treatment, the clinical results from these patients are observed and described.

* Group 1 (Simpson stage 1-3): Beginning no later than 6 weeks following surgery, patients undergo radiotherapy once daily, 5 days a week for 6 weeks.
* Group 2 (Simpson stage 4-5): Beginning no later than 6 weeks following surgery, patients undergo radiotherapy once daily, 5 days a week for 7 weeks.

Patients complete a Mini-Mental Status Exam at baseline and at 6 weeks and 6 months after completion of study.

After completion of study treatment, patients are followed at 6 weeks, at 6 and 12 months, and then annually for at least 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed meningioma, including the following subtypes:

  * Atypical WHO grade II meningioma greater than or equal to 4 mitosis per high-power field [HPF] or the presence of at least 3 of the following variables:

    * Cellularity
    * Architectural sheeting (i.e., patternless pattern)
    * Macronuclei cell formation
    * Small cell formation
  * Malignant WHO grade III meningioma
* All locations allowed except for optic nerve sheets tumors
* Complete or subtotal resection as assessed by the surgeon after verification with a postoperative MRI and according to Simpson guidelines
* No neurofibromatosis type 2 (NF-2)

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Not pregnant or nursing
* Fertile patients must use effective contraception during study therapy
* May be registered on this trial only once
* No clinical evidence of second malignancies except carcinoma in situ of the cervix or basocellular carcinoma
* No psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol and follow-up schedule

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy to the brain or meninges interfering with the protocol treatment plan

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Adverse events as assessed by NCI CTCAE v3.0
Mini-mental status exam
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Damien C. Weber, MD, PhD, Study Chair — Hopital Cantonal Universitaire de Geneve
Locations (1):
- Hopital Cantonal Universitaire de Geneve, Geneva, Switzerland